CLINICAL TRIAL: NCT04177485
Title: Evaluating a Caregiver SMS Reminder Intervention to Reduce Immunization Drop-out in Arua, Uganda-a Randomized Controlled Trial
Brief Title: Evaluating a Caregiver SMS Reminder Intervention to Reduce Immunization Drop-out in Arua, Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: African Field Epidemiology Network (Unknown); Ministry of Health, Uganda (Other Government); Health Information Systems Programme-Uganda (Unknown); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Daniel Ehlman, Principal Investigator, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6721
Record Dates: First submitted 2019-11-05; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Diphtheria; Tetanus; Pertussis; Polio; Measles; Hepatitis B; Haemophilus Influenzae Type b Infection
Keywords: SMS reminder; vaccination; immunization; vaccination drop-out; vaccination timeliness; text reminder; mHealth; cell phone; mobile phone
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis; Measles; Hepatitis B; Haemophilus Infections

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care + SMS text reminders (Experimental): Standard of Care + SMS text reminders to be sent to caregivers for each of their subsequent vaccination visits, as per the EPI schedule (Penta2/OPV2/PCV2, Penta3/OPV3/PCV3, and MCV)
  Interventions: Behavioral: SMS text reminders
- Standard of Care (No Intervention): *Standard of care was defined as the health worker providing vaccination cards (home based records) to caregivers, as available, and providing verbal instruction of when to return for the next visit.

INTERVENTIONS:
Behavioral: SMS text reminders — SMS reminders (in English and the local language) for the 2nd dose of Pentavalent vaccine were sent 28, 30 and 32 days after the 1st dose. SMS reminders for the 3rd dose of Pentavalent vaccine were sent 61, 66, and 68 days after the 1st dose. SMS reminders for the measles-containing vaccine were sent 274, 279, and 281 days after the child's date of birth.
  Arms: Standard of Care + SMS text reminders

SUMMARY:
Faced with high rates of immunization drop-out, Uganda's immunization program requires innovative approaches to address this weakness. Building upon Uganda's growing mHealth infrastructure to pilot a scalable short message service (SMS) system to remind caregivers of their children's upcoming vaccination visits, it was hypothesized that the SMS intervention will increase immunization coverage in a cost-effective and affordable manner that would make it scalable. The study design was an investigator-blinded, multi-center, parallel groups randomized controlled trial with randomization occurring at the caregiver level in select health facilities of Arua District in Uganda. Enrollment took place at the time of Pentavalent 1 vaccination, and both arms included standard of care provided by the health worker. However, in the intervention arm, caregivers also received SMS text messages reminding them to return for their children's second and third doses of Pentavalent vaccine (four and eight weeks after the first dose of Pentavalent vaccine) and measles-containing vaccine (9 months of age). The primary outcome of interest is vaccination coverage at 12 months of age among children enrolled in the study and will be measured by comparing Penta3 and MCV coverage between arms. The study will also examine the SMS impact on timeliness of vaccine receipt, as it is hypothesized that those children receiving the SMS intervention will be more likely to have timely vaccination than those in the control group. The study will also assess caregiver acceptability and cost-effectiveness of the SMS intervention. In addition to assessing its impact on strengthening the immunization program, this intervention has implications for strengthening other programs of the health system through similar health messaging directed toward caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Is a caregiver of a child between the ages of 6 weeks and 6 months of age and presents at one of the study sites for child's Penta1 vaccination
* Access to a personal or household cell phone that can receive text messages
* Lives in Arua district

Exclusion Criteria:

* Does not have access to the cell phone number at time of registration
* Does not agree or is unable to consent to participate in the study
* Does not anticipate being the caregiver through the child's first birthday
* Plans to move out of Arua district in the upcoming year
* Prior enrollment of the caregiver with a different child

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1962 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Number of participants who received MCV by 12 months of age as assessed by data abstraction of home-based records at endline survey. | through study completion, an average of 12 months in the study

SECONDARY OUTCOMES:
Number of participants who received all eligible vaccines (Penta2, PCV2, Polio2, Penta3, PCV3, Polio3, MCV) as assessed by data abstraction of home-based records and caregiver recall at endline survey. | through study completion, an average of 12 months in the study
Number of participants who received Penta3 within 12 weeks of Penta1 as assessed by data abstraction of home-based records at endline survey. | through study completion, an average of 12 months in the study
Number of participants who received MCV by 10 months of age as assessed by data abstraction of home-based records at endline survey. | through study completion, an average of 12 months in the study
Number of participants who would be interested in receiving SMS immunization reminders for their next child, as assessed with a yes/no question at the endline survey. | through study completion, an average of 12 months in the study
Cost per additional child that is up-to-date with vaccination | through study completion, an average of 12 months in the study
  From the MOH perspective, what is the cost-effectiveness of the SMS reminder system per additional child that is up-to-date with vaccination?
Number of participants who received Penta3 by 12 months of age as assessed by data abstraction of home-based records at endline survey. | through study completion, an average of 12 months in the study

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Ehlman, MPH, Principal Investigator — Centers for Disease Control and Prevention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ehlman DC, Magoola J, Tanifum P, Wallace AS, Behumbiize P, Mayanja R, Luzze H, Yukich J, Daniels D, Mugenyi K, Baryarama F, Ayebazibwe N, Conklin L. Evaluating a Mobile Phone-Delivered Text Message Reminder Intervention to Reduce Infant Vaccination Dropout in Arua, Uganda: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Feb 24;10(2):e17262. doi: 10.2196/17262. PMID 33625372